CLINICAL TRIAL: NCT06688799
Title: A Single-Center, Open-Label, Non-Randomized, Single-Arm Clinical Study on the Treatment of Refractory Autoimmune Diseases With CD19-CAR T Cells
Brief Title: Anti-CD19 Chimeric Antigen Receptor T Cells for Refractory Autoimmune Diseases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Principal Investigator, Jing Pan, Director of Dept of Hemato-Oncology and Immunotherapy, Beijing GoBroad Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BJGBYY-IIT-LCYJ-2024-046
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Autoimmune Diseases
Keywords: Refractory Autoimmune Diseases; CD19 CAR-T
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental : CD19 CAR (Experimental): Following the lymphodepleting treatment, patients will be treated with CD19 Chimeric Antigen Receptor (CAR) positive T cells as a single dose.
  Interventions: Drug: CD19 CAR-T cells

INTERVENTIONS:
Drug: CD19 CAR-T cells — Following lymphodepletion with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with CD19 Chimeric Antigen Receptor (CAR) positive T cells as a single dose.

SUMMARY:
The goal of this study is to evaluate the safety and effi cacy of CD19 CAR T cells in the treatment of Refractory Autoimmune Diseases.

DETAILED DESCRIPTION:
This is a single-center, open-label, non-randomized, Phase I/II trial. Patients with Refractory Autoimmune Diseases will receive CD19 CAR T cells. The primary objective is to learn about the safety and tolerability of CD19 CAR T cell therapy in subjects with Refractory Autoimmune Diseases and to determine the optimal biological dose (OBD) and recommend phase 2 dose (RP2D) in phase I and to learn about the efficacy CD19 CAR T-cell therapy in patients with Refractory Autoimmune Diseases in phase II. The primary endpoint is type and incidence of dose limiting toxicity (DLT) within 28 days after CD19 CAR T-cell infusion in phase I and overall response rate (ORR) in phase II. A total number of 18 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Systemic lupus erythematosus (SLE) 1.1. Refractory systemic lupus erythematosus (SLE) and / or refractory lupus nephritis (LN)

1. Male or female patients, aged 3-65 years (including 3 and 65 years);
2. Systemic lupus erythematosus that meets the 2019 American Society of Rheumatology (ACR) / European Association of Rheumatology Consortium (EULAR) classification criteria (see Annex 2);
3. Nuclear antibody (ANA) test is clearly positive, namely ANA titer 1:80 (based on the equivalent results of Hep-2 immunofluorescence or enzyme immunoassay) and / or the test at the screening visit (based on ELISA test, 30 IU / mL).
4. Refractory systemic lupus erythematosus (SLE) and / or refractory lupus nephritis (LN):

<!-- -->

1. Patients take at least 7.5 mg of prednisolone daily to maintain low disease activity or a SLEDAI 2K score (see attachment 3) of 8 or higher.
2. Recurrence of disease activity after failure of conventional therapy or after remission. Definition of conventional treatment: using corticosteroids (1 mg / kg / day) and cyclophosphamide for 6 months; or any of the following immunomodulatory drugs for more than 3 months: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, and biological agents such as rituximab, belimumab, and teacept.

5) Physical strength status score (ECOG): 0-2 points; 6) The estimated survival period of 90 days; 1.2. Immune thrombocytopenia in refractory lupus (SLE-ITP)

1. Age range: 18-70 years (including 18 and 70 years), gender limitation.
2. Patients with refractory systemic lupus erythematosus (immune thrombocytopenia): meeting SLE 2019 ACR / EULAR classification criteria, with at least 2 consecutive routine blood tests showing platelets lower ; no abnormal morphology of blood cells in peripheral blood smear; morphological characteristics of bone marrow cells meeting immune thrombocytopenia. Refractory systemic lupus erythematosus (immune thrombocytopenia) was defined as at least 1 course of MP shock (1g 3 days) or high-dose hormone (1mg / kg d equivalent dose of glucocorticoid) combined with 1 or more immunosuppressive agents. Thrombocytopenia except for other than non-SLE causes, such as infection, myelosuppression, macropleic, hypersplenism, etc.
3. Clinician assessment of the patients condition allowed the use of 10mg prednisone or its equivalent dose during the study and allowed the discontinuation of all immunosuppressive agents (excluding hydroxychloroquine).

   1.3. refractory lupus thrombotic microangiopathy (SLE-TMA)

<!-- -->

1. Age range: 18-70 years (including 18 and 70 years), gender limitation.
2. Meet SLE-TMA standard; meet one of the following criteria, associated with SLE Microvascular hemolytic anemia, associated with elevated lactate dehydrogenase and peripheral blood smear fragmentation; and thrombocytopenia, except for other reasons; Renal biopsy suggested a TMA.

Refractory systemic lupus erythematosus was defined as no TMA response with at least 1 course of MP shock (1g 3 days) or high-dose hormone (1mg / kg d equivalent dose glucocorticoid) combined with 1 or more immunosuppressants.

The clinician assessed the patients condition allowed a glucocorticoid dose of up to 10mg prednisone or its equivalent dose during the study and allowed discontinuation of all immunosuppressive agents (excluding hydroxychloroquine).

1.4.SLE Myelitis

1. Age: 18-60 years old.
2. Diagnosis: meet the diagnostic criteria for SLE.
3. Myelitis: acute or subacute paraplegia, sensory plane, sphincter dysfunction, and tendon reflex or plantar reflex abnormalities; including but not limited to spinal cord lesions confirmed by MRI. And other causes of myelitis.
4. Severity: lower limb muscle strength grade 3
5. Refractory / recurrent nature:

Refractory: ineffective against high-dose hormone shock therapy and / or combined with other immunosuppressants; Relapse: at least two recurrences in the past 12 months, or three times in the past 24 months, and one recurrence in the 12 months prior to screening.

1.5.SLE Pulmonary arterial hypertension (SLE-PAH)

1. Age range: 18-70 years (including 18 and 70 years), gender is unlimited.
2. Patients with refractory connective tissue disease (pulmonary arterial hypertension):

<!-- -->

1. confirmed as systemic lupus erythematosus according to the 1997 ACR or EULAR / ACR revision standard in 2019;
2. meeting the diagnostic criteria for PAH confirmed by a right heart catheter (as defined by 2022 ESC / ERS guidelines for the treatment of pulmonary hypertension): 1) mean pulmonary artery pressure (mPAP) 20mmHg at rest; 2) pulmonary vascular wedge pressure (PAWP) 15mmHg,and pulmonary vascular resistance (PVR)> 2 WUs at rest;
3. PAH did not reach risk stratification for patients in the low-risk group. Low-risk patients need to meet: 1) WHO cardiac function grades I-II; 2) 6 min walking distance (6 MWD)> 440 m; 3) BNP <50 ng/L, or NT-proBNP <300 ng/L; 4) right atrial pressure (RAP) <8mmHg and heart index (CI) 2.5 L · min 1 · m 2.
4. Subjects had received a standard dose of treatment before the first dose of study drug, including glucocorticoids (prednisone 0-30mg / day, or other equivalent) for at least 4 weeks; antimalarials, single-agent immunosuppressors (allowed to apply immunosuppressors limited to: mycophenol ester or mycophenolic acid 1.5g / day, azathioprine or 6-mercaptopurine 2mg / kg / day, methotrexate 15mg / week, leflunomide 20mg / day) for at least 12 weeks and not increased or replaced within 24 weeks after medication. Less than three (including prostaglandin analogues, endothelin receptor, antagonists, PDE-5 inhibitors, guanylate cyclase agonists) and have been stable for at least 4 weeks and do not increase or change within 24 weeks after drug treatment.
5. Clinician assessment of the patients condition allowed the use of glucocorticoids not to 10mg prednisone or its equivalent dose during the study and allowed the withdrawal of all immunosuppressive agents (excluding hydroxychloroquine).

1.6.SLE-Protein loss enteropathy (SLE-PLE)

1. Age range: 18-70 years (including 18 and 70 years).
2. Refractory SLE-PLE:

<!-- -->

1. confirmed as systemic lupus erythematosus according to the 1997 ACR or EULAR / ACR revision standard in 2019;
2. Meet the SLE-PLE standard: meet one of the following standards. Clinical symptoms and laboratory findings associated with PLE, including hypoalbuminemia (urinary protein loss, severe liver disease or malnutrition, which is not completely explained by other pathological mechanisms) Refractory systemic lupus erythematosus was defined as no PLE response after at least 1 course of MP shock (1g 3 days) or high-dose hormone (1mg / kg d equivalent dose of glucocorticoids) combined with 1 or more immunosuppressants.

The clinician assessed the patients condition allowed a glucocorticoid dose of up to 10mg prednisone or its equivalent dose during the study and allowed discontinuation of all immunosuppressive agents (excluding hydroxychloroquine).

（3）Blood pregnancy tests were negative for women of reproductive age within 7 days before trial pretreatment; any fertile male and female patient must agree to effective contraception throughout the study and for at least 2 years. According to the researchers, a patient with fertility means a biological ability to have a living baby and a normal sexual life. Female patients without fertility (i. e., meet at least one following criteria): hysterectomy or bilateral oophorectomy, or medical confirmation of ovarian failure, or postmenopause (at least 12 consecutive months of menopause in the absence of pathological or physiological causes).

2. Sjogrens Syndrome (SS) 2.1.SS-ITP

1. The age at screening was 18 ~ 65 years old (including 18 and 65 years old);
2. Classification classification of primary Sjogrens Syndrome according to the 2002 International Classification or ACR / EULAR in 2016, the diagnosis of primary Sjogrens syndrome for at least 6 months;
3. Positive antinuclear antibody (titer 1:80) at screening, and / or anti-SSA antibody, and / or anti-SSB antibody;
4. Active relapse / refractory SS should meet at least one of the following scenarios:
5. Relapse / refractory immune thrombocytopenia: refractory to first-line therapy, platelet-inducing drugs in second-line therapy and / or rituximab therapy / hormone dependence or intolerance, platelet <30109 / L, and PGA> 1.

2.2.SS Myelitis

1. Age: 18-60 years old.
2. Diagnosis: Meet the diagnostic criteria for Sjogrens syndrome (SS) (such as the American College of Rheumatology (ACR) criteria).
3. The diagnosis of NMOSD requires neurological evaluation and MRI imaging confirmation, meeting the NMOSD diagnostic criteria as follows:

   The NMOSD diagnostic criteria for AQP 4-IgG positivity; At least 1 core clinical feature; AQP 4-IgG using the best available assay.
4. Severity: lower limb muscle strength grade 3
5. Infractability and recurrence:

Refractory: ineffective against high-dose hormone shock therapy and / or combined with other immunosuppressants; Relapse: at least two recurrences in the past 12 months or three in the past 24 months and one in the 12 months prior to screening.

2.3.SS-PAH

1）Age range: 18-70 years (including 18 and 70 years), gender is unlimited. 2）Patients with refractory connective tissue disease (pulmonary arterial hypertension):

1. Meet the 2002 AECG classification criteria or 2016 ACR / EULAR classification criteria, and diagnosed as primary Sjogrens syndrome;
2. meeting the diagnostic criteria for PAH confirmed by a right heart catheter (as defined by the 2022 ESC / ERS guidelines for the treatment of pulmonary hypertension): 1) mean pulmonary artery pressure (mPAP) 20mmHg at rest; 2) pulmonary vascular wedge pressure (PAWP) 15mmHg; and pulmonary vascular resistance (PVR)> 2 WUs at rest;
3. PAH did not reach risk stratification for patients in the low-risk group. Low-risk patients need to meet: 1) WHO cardiac function grades I-II; 2) 6 min walking distance (6 MWD)> 440 m; 3) BNP <50 ng/L, or NT-proBNP <300 ng/L; 4) right atrial pressure (RAP) <8mmHg and heart index (CI) 2.5 L · min 1 · m 2.
4. Subjects had received a standard dose of treatment before the first dose of study drug, including glucocorticoids (prednisone 0-30mg / day, or other equivalent) for at least 4 weeks; antimalarials, single-agent immunosuppressors (allowed to apply immunosuppressors limited to: mycophenol ester or mycophenolic acid 1.5g / day, azathioprine or 6-mercaptopurine 2mg / kg / day, methotrexate 15mg / week, leflunomide 20mg / day) for at least 12 weeks and not increased or replaced within 24 weeks after medication. Less than three (including prostaglandin analogues, endothelin receptor, antagonists, PDE-5 inhibitors, guanylate cyclase agonists) and have been stable for at least 4 weeks and do not increase or change within 24 weeks after drug treatment.
5. Clinician assessment of the patients condition allowed the use of glucocorticoids not to 10mg prednisone or its equivalent dose during the study and allowed the withdrawal of all immunosuppressive agents (excluding hydroxychloroquine).

3. Systemic sclerosis (SSc) 3.1.SSc-ILD And skin sclerosis

1. the diagnosis of SSc was confirmed according to the 2013 ACR / EULAR classification criteria
2. Course of disease for 6 years after the first presentation of non-Raynaud phenomenon
3. Age is 18 years old, 70 years old, gender is not limited in patients with ILD (1) ILD confirmed by chest HRCT, range 20%, ground glass shadow or grid shadow (2) Lung function: FVC% 60%, and DLCO 40% (3) MMF or CTX for more than 3 months (shortness of breath aggravation, or 5% decrease in FVC% or 10% decrease in DLCO%, or chest HRCT aggravation, except for infection and other factors)
4. Skin sclerosis:

(1) Patients with dcSSc (2) mRSS 12 points, or new skin involvement areas or skin progression (mRSS 3 points) were recorded in the past 6 months (3) Previous application of hormones / immunosuppressants / JAK inhibitors / biological agents has poor efficacy 3.2.SSc-PAH

1)Age range: 18-70 years (including 18 and 70 years), gender is unlimited. 2)Patients with refractory connective tissue disease (pulmonary arterial hypertension):

1. Meet the 1980 ACR or ACR / EULAR classification criteria in 2013 and make a diagnosis of systemic sclerosis.
2. meeting the diagnostic criteria for PAH confirmed by a right heart catheter (as defined by the 2022 ESC / ERS guidelines for the treatment of pulmonary hypertension): 1) mean pulmonary artery pressure (mPAP) 20mmHg at rest; 2) pulmonary vascular wedge pressure (PAWP) 15mmHg; 3) and pulmonary vascular resistance (PVR)> 2 WUs at rest;
3. PAH did not achieve risk stratification for patients in the low-risk group. Low-risk patients need to meet: 1) WHO cardiac function grades I-II; 2) 6 min walking distance (6 MWD)> 440 m; 3) BNP <50 ng/L, or NT-proBNP <300 ng/L; 4) right atrial pressure (RAP) <8mmHg and heart index (CI) 2.5 L · min 1 · m 2.
4. Subjects had received a standard dose of stable treatment before the first dose of study drug, including glucocorticoids (prednisone 0-30mg / day, or equivalent) for at least 4 weeks; antimalarials, single-agent immunosuppressive agents (limited to moxachenolate or mycophenolic acid 1.5g / day, azathioprine or 6-mercaptopurine 2mg / kg / day, methotrexate 15mg / week, leflunomide 20mg / day) for at least 12 weeks and not increased or replaced within 24 weeks after treatment. Less than three (including prostaglandin analogues, endothelin receptor, antagonists, PDE-5 inhibitors, guanylate cyclase agonists) and have been stable for at least 4 weeks and do not increase or change within 24 weeks after drug treatment.
5. Clinician assessment of the patients condition allowed the use of glucocorticoids not to 10mg prednisone or its equivalent dose during the study and allowed the withdrawal of all immunosuppressive agents (excluding hydroxychloroquine).

4. Antiphospholipid syndrome (APS)

1. Selected patients or their legal representatives shall voluntarily sign the informed consent form.
2. Age range: 18-70 years (including 18 and 70 years), gender is unlimited.
3. Patients with refractory APS (immune thrombocytopenia, microangiopathic APS): APS with microangiopathy and / or immune thrombocytopenia (APS-ITP).

Patients with refractory microangiopathic APS: according to the 2023 ACR / EULAR classification criteria for APS nephropathy, myocardial lesions, alveolar hemorrhage, adrenal hemorrhage or microthrombosis, or meet the 2003 CAPS classification criteria. Refractory APS was defined as a shock to corticosteroids or high-dose hormone combined with at least one immunosuppressive agent (including CTX, tacrolimus, MMF and cyclosporin) induced remission for 3 months with continued progression or no resolution of microangiopathy.

Patients with refractory APS-ITP: at least 2 consecutive routine blood tests showed platelets lower than 50109 / L; microscopic morphology of blood cells in peripheral blood smear; morphological characteristics of bone marrow cells were immune thrombocytopenia. Refractory APS-ITP (immune thrombocytopenia) was defined as receiving at least 1 course of MP shock (1g 3 days) or a high dose of hormone (1mg / kg d equivalent dose of glucocorticoid) combined with 1 or more immunosuppressive agents did not achieve at least partial response. Except thrombocytopenia other non-APS causes, such as infection, bone marrow suppression, macropleism and hypersplenism.

The clinician assessed the patients condition allowed a glucocorticoid dose of up to 10mg prednisone or its equivalent dose during the study and allowed discontinuation of all immunosuppressive agents (excluding hydroxychloroquine).

5. Idiopathic inflammatory myopathy (IIM)

1. Age range: 1870 years (including 18 and 70 years), gender unlimited, weight 40 kg at screening.
2. Classification criteria: IIM patients: must meet the "positive" or "very likely" diagnosis (Lundberg et al 2017) according to the EULAR / ACR adult idiopathic inflammatory myopathy (IIM) classification criteria, or by the 2010 Connors et al.
3. Definition of refractory IIM: at least one immunosuppressive agent (e. g., azathioprine, methotrexate, mycophenolate, cyclosporine, tacrolimus, cyclohamide, leflunomide, etc.) that has received stable doses for over 2 months, When corticosteroids were reduced to 10mg daily prednisone or its equivalent dose or above, At least one of the following deterioration occurred: (i) ILD progression, The symptoms of shortness of breath worsened after the activity, Or an increased ILD score for lung HRCT, Or pulmonary function FVC% predicted decrease greater than 5%, Or DLco% decrease of> 10%; And (ii) deterioration of myositis, MMT-8 decreased> 5 points / 150 points, Or creatine kinase elevated> 100U / L.
4. Definition of recurrent IIM: The reappearance of active IIM after 6 months of sustained disease remission causes new organ involvement or aggravation of the original involved organ, or the need for increased glucocorticoids and immunosuppressive agents.
5. The clinician assessing the patients condition allowed the use of glucocorticoid doses not exceeding 10mg prednisone or its equivalent dose during the study period and permitted the discontinuation of all immunosuppressants.

6. Anti-neutrophil cytoplasic antibody-associated vasculitis (AAV: GP A/MPA)

1. Severe patients diagnosed with GPA or MPA according to 2022 ACR / EULAR criteria, treated with cyclophosphamide or hormone with rituximab (BVAS score of 0), or relapsed with maintenance therapy with rituximab or cyclophosphamide.(Recurrence is defined as the occurrence of at least one primary item, or 3 secondary items, or an abnormality of 1 or 2 secondary items in two consecutive follow-ups);
2. The patient is positive for ANCA (anti-MPO or PR3 antibody) at present or during the course of the disease.

   Exclusion Criteria: An individual who meets any of the following criteria will be excluded from participation in this study:

1. intracranial hypertension or cerebral consciousness disorder: Intracranial pressure is kept above 15mmHg; Organic encephalopathy syndrome, cerebrovascular accident, encephalitis or central nervous system vasculitis, visual impairment and other brain lesions that require intervention.

2. Symptomatic heart failure or severe arrhythmia: Left ventricular ejection fraction (LVEF) <45% within 12 months prior to screening; Abnormal electrocardiogram (ECG): left bundle branch, double bundle branch block or other clinically significant abnormal electrocardiogram; Congenital long QT interval (QT) syndrome or Fridericia correction formula (QTcF) 470 ms; Congestive heart failure (New York Heart Association Class III or IV); 3. Severe respiratory failure or other respiratory symptoms that are difficult to control: 4. Along with other types of malignant tumors; 5. Diffuse endovascular coagulation; 6. Sepsis or other infections that are difficult to control: uncontrolled active systemic bacterial, viral, fungal or parasitic infections (except nail fungal infections) or other clinically significant active diseases; 7. Uncontrolled diabetes: fasting blood glucose (FBG)≥8.0mmol/L, 2 hours postprandial blood glucose (PBG) 15 mmol/L, glycated hemoglobin (HbA 1 c) after at least 3 months of diet, exercise or related treatment; combined with diabetic ketoacidosis or other uncontrollable diabetic complications; 8. Received organ transplantation (excluding bone marrow transplantation); 9. eGFR CKD-EPI < 30 ml/min/1.73m^2； 10. Patients who cannot continue the immunosuppressive agents for 7 days, or repeat the disease and the investigators evaluate the risk of serious adverse reactions.

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-23 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Phase I:Dose-limiting toxicity (DLT) | 28 days post infusion
  The incidence and type of dose-limiting toxicity (DLT).
Phase I： Adverse events (AEs) | 30 days post infusion
  The incidence and severity of adverse events (AE).
Phase II: Objective response rate (ORR) | 3 months and 6 months post infusion]
  Proportions of subjects achieving Autoimmune Diseases response

SECONDARY OUTCOMES:
Phase I: Objective response rate (ORR) | 3 months and 6 months
  Proportions of subjects achieving Autoimmune Diseases response.
Phase I: Long-term serious adverse events (SAEs) | From 30 days after CD19 CAR T infusion to 2 years
  Total number, incidence and severity of SAEs from 30 days to 2 years after CD19 CAR T infusion will be recorded.
Phase I: Pharmacokinetics(PK) | Up to 2 years post infusion
  The proliferation and survival of CD19 CAR T cells will be measured by flow cytometry and quantitative polymerase chain reaction (qPCR).
Phase I: Pharmacodynamic(PD) | Up to 2 years post infusion
  The lymphocyte Subsets Detection and cytokine Detection will be measured by flow cytometry.
Phase II: Adverse events (AEs) | 2 years post infusion
  The incidence and severity of adverse events.
Phase II: Pharmacokinetics（PK） | Up to 2 years post infusion
  The proliferation and survival of CD19 CAR T cells will be measured by flow cytometry and quantitative polymerase chain reaction (qPCR).
Phase II: Pharmacodynamic(PD) | Up to 2 years post infusion
  The lymphocyte Subsets Detection and cytokine Detection will be measured by flow cytometry.
Phase II: Overall survival (OS) | Up to 2 years post infusion
  Overall survival (OS) is defined the time from the initial CD19 CAR T cell infusion to death for any cause.
Phase II:During of response (DOR) | Up to 2 years post infusion
  During of response (DOR) is defined as the date when response criteria are first met to the date of relapse or death caused by Autoimmune Diseases in the absence of documented relapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing GoBroad Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No